CLINICAL TRIAL: NCT00912067
Title: Ocular Graft Versus Host Disease After Hematopoietic Stem Cell Transplantation in Adults
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Irina Barequet MD/PI, Sheba Medical Center
Other Study IDs: SHEBA-09-7085-IB-CTIL
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hematopoietic stem cell transplantation

SUMMARY:
The purpose of this study is to evaluate the presence and manifestations of ocular graft versus host disease in adults that had hematopoietic stem cell transplantation in the past 3 years at the sheba medical center, Israel. As well as correlate the degree of the presentation to the therapeutic protocol (chemotherapy and irradiation).

ELIGIBILITY:
Inclusion Criteria:

* after hematopoietic stem cell transplantation done at sheba medical center Israel
* 3 month have past from transplantation but no more then 3 years

Exclusion Criteria:

* transplantation done in the last 3 month or more than 3 years have past since

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults after hematopoietic stem cell transplantation done at sheba medical center Israel during the last 3 years
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-07

CONTACTS AND LOCATIONS:
Overall Officials: irina barequet, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Kim SK. Update on ocular graft versus host disease. Curr Opin Ophthalmol. 2006 Aug;17(4):344-8. doi: 10.1097/01.icu.0000233952.09595.d8. PMID 16900025
- [Background] Anderson NG, Regillo C. Ocular manifestations of graft versus host disease. Curr Opin Ophthalmol. 2004 Dec;15(6):503-7. doi: 10.1097/01.icu.0000143684.22362.46. PMID 15523196